CLINICAL TRIAL: NCT04962061
Title: Impacts of Aerobic, Resistance and Cognitive Training Interventions on Neurocognitive Functions in Older Adults With Cardiovascular Risk Factors.
Brief Title: A Combined Multidomain Intervention to Prevent Cognitive Decline Associated With Cardiovascular Risk Factors.
Acronym: ACTIONcR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Bherer (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Montreal Health Innovations Coordinating Center (MHICC) (Other)
Responsible Party: Sponsor-Investigator, Louis Bherer, Director of the EPIC Center and Scientist, Montreal Heart Institute, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-2545
Record Dates: First submitted 2021-06-16; First posted 2021-07-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Aging; Cardiovascular Risk Factor
Keywords: Aging; Cardiovascular Risk factor; Cognition; Combined Intervention; Cognitive Training; Physical Exercise; Brain Functions; Biomarkers
MeSH Terms: conditions — Motor Activity | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This clinical trial is a double-blinded study. Research personnel performing the outcome assessments will be blinded to group allocation. Participants will be aware of the type of training they receive, but they will be blinded to the "active" intervention and study hypotheses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Multidomain intervention (Experimental): The multidomain intervention will combine a cognitive training with aerobic and resistance exercises training, three sessions per week for 46 weeks. Participants will be allowed to perform cognitive and exercise training sessions either home-based or centre-based.
  Interventions: Other: Cognitive Training; Other: Aerobic and resistance exercises
- Physical exercise intervention (Experimental): The physical exercises intervention will include aerobic and resistance exercises training, three sessions per week for 46 weeks. Participants will be allowed to perform cognitive and exercise training sessions either home-based or centre-based.
  Interventions: Other: Aerobic and resistance exercises
- Active control intervention (Active Comparator): The active control intervention will include stretching and toning exercises, three sessions per week for 46 weeks. Participants will be allowed to perform cognitive and exercise training sessions either home-based or centre-based.
  Interventions: Other: Stretching and Toning

INTERVENTIONS:
Other: Cognitive Training — Participants will be encouraged to perform sessions of cognitive training 3 times per week (30 minutes/session). Two of these sessions will involve computer- or tablet-based attentional control training targeting dual-tasking, updating and working memory, as well as inhibition and switching. Difficulty of cognitive training will be tailored to participants' performances. The remaining session will consist of memory training. Participants will be instructed mnemotechnic, as well as be taught about memory in aging in general.
  Arms: Multidomain intervention
Other: Aerobic and resistance exercises — Participants will follow a periodized exercise training program with thrice-weekly 60 minutes trainings. The sessions will start with a 5-10mins warm-up, followed by aerobic and resistance trainings, and ends with a 5-10mins cool-down and stretching period. Intensity of aerobic sessions will be monitored with heart rate chest strap and should match with the moderate to vigorous intensity zone as defined by the ACSM (65% of Heart Rate maximum or more and a Perceived Exertion higher than 12 on the 6 to 20 Borg scale). Exercise intensity and duration will be gradually increased during the program. After aerobic training, a 15-20mins resistance training will be performed with a gradual progression of higher intensities and/or numbers of sets. The one maximal repetition (1RM) will be assessed for each RT movements at baseline, during (each 3 months) and at the end of the program. RT intensities will go from 40 to 70% of 1RM, with 8 to 10 forms of exercise involving majors muscle groups.
  Arms: Multidomain intervention; Physical exercise intervention
Other: Stretching and Toning — Participants in the active control condition will take part in three 60 minutes stretching and toning sessions per week. Each session will start with a five-minutes warm-up, followed by fifteen min of body stretching exercises mainly in a seated position and finish with a five-minutes cool down. Participants will engage in four muscle-toning exercises (light intensity) using dumbbells or resistance bands, two exercises designed to improve balance, one yoga sequence, and one exercise of their choice. Intensity of stretching and toning sessions will be monitored with heart rate chest strap and should not exceed the light intensity zone as defined by the ACSM (64% of Heart Rate maximum or less and a Perceived Exertion lower than 11 on the 6 to 20 Borg scale).
  Arms: Active control intervention

SUMMARY:
The ACTIONcardioRisk trial is designed to investigate the effect of aerobic and progressive resistance training exercises combined with cognitive training, on neurocognitive functioning of sedentary older adults with and without cardiovascular risk factors.

DETAILED DESCRIPTION:
The proportion of older adults is on the rise in Canada, with the fastest growth recorded among those seventy years of age or older. The prevalence of cardiovascular risk factors (CVRF) such as diabetes, hypertension, and high cholesterol increases drastically with age. Individuals with CVRF often show impaired cognition, such as attention and memory deficits. In healthy older adults, exercise training and cognitive stimulation can help enhance cognitive performances. More precisely, combined intervention, including physical and cognitive training, has shown beneficial effects on cognition in older adults without cognitive impairment and with mild cognitive impairment. However, the effect of such programs on cognition in individuals with CVRF is not well documented. This project compares the effect of a physical exercise program, including aerobic and resistance training, alone or combined with cognitive training on cognitive performances and brain imaging outcomes in individuals with CVRF and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 60 and older,
* Normal or corrected vision and normal hearing for their age range,
* No cognitive impairment (Mini-Mental State Examination - MMSE ≥ 25),
* Inactive (< 150 min of physical activity per week).

Exclusion Criteria:

* MMSE ≤ 24 or diagnosis of dementia,
* Uncontrolled psychological / psychiatric condition within the past 6 months,
* Neurological disease,
* Severe exercise intolerance,
* Respiratory disease (e.g., asthma, COPD),
* Excessive alcohol consumption (> 15 drinks/week),
* Documented cerebral, peripheral or coronary atherosclerotic disease,
* Chronic systolic or diastolic heart failure,
* Symptomatic aortic stenosis,
* Atrial fibrillation,
* Automatic implantable defibrillator or permanent pacemaker,
* Malignant exertional arrhythmias,
* Non-cardiopulmonary limitation to exercise (e.g., arthritis).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in general cognitive functioning | Baseline and post-intervention at 12 months.
  Montreal Cognitive Assessment (0-30 score, with a higher score indicating a better cognitive functioning).
Change in processing speed | Baseline and post-intervention at 12 months.
  Validated remote version of neuropsychological tests and iPad tests (Composite Z-score).
Change in executive functions | Baseline and post-intervention at 12 months.
  Validated remote version of neuropsychological tests and iPad tests (Composite Z-score).
Change in episodic memory | Baseline and post-intervention at 12 months.
  Validated remote version of neuropsychological tests and iPad tests (Composite Z-score).

SECONDARY OUTCOMES:
Change in cerebral autoregulation - frontal cortical region | Baseline and post-intervention at 12 months.
  Variations of prefrontal cortical oxygen saturation (rSO2, [HbO]/([HbO]+[HbR])) will be measured by Near Infrared Spectroscopy (NIRS), as a surrogate of cortical blood flow. Variations of continuous peripheral blood pressure (mm Hg) will be simultaneously measured by plethysmography at the finger. Autoregulation indices (unitless) will be derived from the correlation between variations of oxygen saturation measures and variations of peripheral blood pressure.
Change in cerebral autoregulation - middle cerebral arteries | Baseline and post-intervention at 12 months.
  Variations of cerebral blood flow velocity (cm/s) at the level of the middle cerebral artery will be measured by Transcranial Doppler (TCD). Variations of continuous peripheral blood pressure (mm Hg) will be simultaneously measured by plethysmography at the finger. Autoregulation indices (unitless) will be derived from the correlation between variations of cerebral blood flow measures and variations of peripheral blood pressure.
Change in cerebral vasoreactivity - whole brain | Baseline and post-intervention at 12 months.
  Cerebral VasoReactivity (CVR, % change per mm Hg of PaCO2) will be measured by Arterial Spin Labeling MRI in two third of the study participants who do not present contra-indication for imaging studies.
Change in cerebral vasoreactivity - prefrontal cortex | Baseline and post-intervention at 12 months.
  Cerebral VasoReactivity (CVR, % change per mm Hg of PaCO2) will be measured using NIRS in the prefrontal region.
Change in cerebral vasoreactivity - middle cerebral arteries | Baseline and post-intervention at 12 months.
  Cerebral VasoReactivity (CVR, % change per mm Hg of PaCO2) will be measured using TCD in the middle cerebral arteries
Change in cerebral pulsatility - cortical frontal region | Baseline and post-intervention at 12 months.
  Pulsatility will be measured as the normalized difference of relative near-infrared light intensity changes between systole and diastole, using NIRS in the prefrontal cortical region.
Change in cerebral pulsatility - middle cerebral arteries | Baseline and post-intervention at 12 months.
  Pulsatility will be measured as the normalized difference of relative blood flow velocities between systole and diastole, using TCD in the middle cerebral arteries.
Change in cerebral activity | Baseline and post-intervention at 12 months.
  Significant changes in brain activity evoked by a Stroop task relative to baseline will be assessed by t-statistics maps, computed from variations of [HbO] and [HbR] measured by NIRS at the prefrontal cortex.
Change in brain structure | Baseline and post-intervention at 12 months.
  Multimodal structural MRI will be performed in two third of the study participants who do not present contra-indication for imaging studies, to measure regional cerebral volumes, as well as volume of angiopathic markers (eg lacunes, microbleeds, white matter hyperintensities), in cm3.

OTHER OUTCOMES:
Change in cardiorespiratory fitness | Baseline and post-intervention at 12 months.
  Maximum incremental cardiopulmonary exercise test (VO2 max (ml.kg.min)).
Change in peripheral endothelial function | Baseline and post-intervention at 12 months.
  Fow-mediated dilation of the brachial artery (%).
Change in central artery stiffness | Baseline and post-intervention at 12 months.
  Carotid femoral pulse-wave velocity (m/s).
Change in walking speed | Baseline and post-intervention at 12 months.
  Timed 10-meter walking test (cm/s).
Change in functional mobility | Baseline and post-intervention at 12 months.
  Timed Time up and Go test (s).
Change in Balance performance | Baseline and post-intervention at 12 months.
  Timed one-leg standing test (s).
Change in lower limb muscles strength | Baseline and post-intervention at 12 months.
  Timed Sit-to-Stand test (s)
Change in upper limb muscle strength | Baseline and post-intervention at 12 months.
  Grip strength test score (kg).
Change in total cholesterol | Baseline and post-intervention at 12 months.
  Total cholesterol levels (mmol/L)
Change in cholesterol-HDL | Baseline and post-intervention at 12 months.
  Cholesterol-HDL levels (mmol/L)
Change in cholesterol-LDL calculated | Baseline and post-intervention at 12 months.
  Cholesterol-LDL calculated levels (mmol/L)
Change in cholesterol non-HDL | Baseline and post-intervention at 12 months.
  Cholesterol non-HDL levels (mmol/L)
Change in triglycerides | Baseline and post-intervention at 12 months.
  Triglycerides levels (mmol/L)
Change in glucose | Baseline and post-intervention at 12 months.
  Glucose levels (mmol/L)
Change in glycated hemoglobin (HbA1c) | Baseline and post-intervention at 12 months.
  Glycated hemoglobin (HbA1c) (%)
Change in insulin | Baseline and post-intervention at 12 months.
  Insulin levels (pmol/L)
Change in creatinine | Baseline and post-intervention at 12 months.
  Creatinine levels (mg/dL)
Change in sodium | Baseline and post-intervention at 12 months.
  Sodium levels (mmol/L)
Change in chloride | Baseline and post-intervention at 12 months.
  Chloride levels (mmol/L)
Change in potassium | Baseline and post-intervention at 12 months.
  Potassium levels (mmol/L)
Change in high-sensitive C-reactive protein (hsCRP) | Baseline and post-intervention at 12 months.
  High-sensitive C-reactive protein (hsCRP) levels (mg/L)
Change in apolipoprotein B (ApoB) | Baseline and post-intervention at 12 months.
  Apolipoprotein B (ApoB) levels (g/L)
Change of neurotrophic biomarkers | Baseline and post-intervention at 12 months.
  Brain-derived neurotrophic factor (BDNF) plasma concentration (pg/mL).
Change in transcriptomics | Baseline and post-intervention at 12 months.
  Transcriptome analysis to assess the impact of the intervention on any changes in the activity of different cellular processes.
Change in gut microbiome | Baseline and post-intervention at 12 months
  DNA extraction from fecal samples. The fecal samples will be collected from the participants who are also performing MRI.
Change in chronic stress levels | Baseline and post-intervention at 12 months.
  Cortisol levels from saliva samples (nmol/L). The saliva samples will be collected from the participants who are also performing MRI.
Change in perceived stress | Baseline and post-intervention at 12 months.
  Perceived Stress Scale questionnaire (Score ranges from 0-4, with 0 no stress,1 mild stress, 3 moderate stress and 4 severe).
Change in anxiety | Baseline and post-intervention at 12 months.
  State-Trait Anxiety Inventory questionnaire (Score ranges from 20-80, with a higher score indicating higher anxiety).
Change in depressive symptoms | Baseline and post-intervention at 12 months.
  Geriatric Depression Scale questionnaire (Score ranges from 0-30, with a higher score indicating larger depressive symptomatology).
Change in health related quality-of-life | Baseline and post-intervention at 12 months.
  12-Item Short Form Health Survey (a completer).
Change in sleep quality | Baseline and post-intervention at 12 months.
  Pittsburg Sleep Quality Index questionnaire (Score ranges from 0-21, with a higher score indicating worse sleep quality).
Change in Dietary patterns | Baseline and post-intervention at 12 months.
  Short Diet Questionnaire (Score ranges from 15-45 points, with a score between 15-29 categorised as unhealthy, 30-37 as somewhat unhealthy, and 38 or more as a healthy diet).
Change in social and community activities involvement | Baseline and post-intervention at 12 months.
  Social and community involvement questionnaire (Score ranges from 0-200, with a higher score indicating more social and community involvement).
Change in self-reported physical activity | Baseline
  Physical Activity Scale for the Elderly questionnaire (Score ranges from 0-400, with a higher score indicating better level of physical activity).
Self-reported masculinity and femininity trait | Baseline
  Short Form Bem Sex-Role Inventory questionnaire (30 items questionnaire with 10 items assessing the femininity traits, 10 items assessing the masculinity traits, and 10 items neutral, not scored. Two scores are calculated for femininity and masculinity, respectively, and range from 10-70, whit a higher score indicating a higher femininity or masculinity trait).
Genetic biomarkers | Baseline
  Genotyping array to generate high quality genome-wide genotyping data that include the APOE and BDNF genes.
Cognitive Reserve | Baseline
  Rami and colleagues' cognitive reserve questionnaire (Scale ranges from 0-26, with a higher score indicating a greater cognitive reserve).
Baseline level of physical activity | Baseline
  Quantification of physical activity using an accelerometry recording of 7 days (minutes of moderate to vigorous activity).

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bherer, PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Preventive medicine and physical activity centre (centre EPIC), Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arntzen KA, Schirmer H, Wilsgaard T, Mathiesen EB. Impact of cardiovascular risk factors on cognitive function: the Tromso study. Eur J Neurol. 2011 May;18(5):737-43. doi: 10.1111/j.1468-1331.2010.03263.x. Epub 2010 Dec 8. PMID 21143340
- [Background] Baker LD, Frank LL, Foster-Schubert K, Green PS, Wilkinson CW, McTiernan A, Cholerton BA, Plymate SR, Fishel MA, Watson GS, Duncan GE, Mehta PD, Craft S. Aerobic exercise improves cognition for older adults with glucose intolerance, a risk factor for Alzheimer's disease. J Alzheimers Dis. 2010;22(2):569-79. doi: 10.3233/JAD-2010-100768. PMID 20847403
- [Background] Bherer L, Kramer AF, Peterson MS, Colcombe S, Erickson K, Becic E. Training effects on dual-task performance: are there age-related differences in plasticity of attentional control? Psychol Aging. 2005 Dec;20(4):695-709. doi: 10.1037/0882-7974.20.4.695. PMID 16420143
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] DeRight J, Jorgensen RS, Cabral MJ. Composite cardiovascular risk scores and neuropsychological functioning: a meta-analytic review. Ann Behav Med. 2015 Jun;49(3):344-57. doi: 10.1007/s12160-014-9681-0. PMID 25616781
- [Background] Dregan A, Stewart R, Gulliford MC. Cardiovascular risk factors and cognitive decline in adults aged 50 and over: a population-based cohort study. Age Ageing. 2013 May;42(3):338-45. doi: 10.1093/ageing/afs166. Epub 2012 Nov 25. PMID 23179255
- [Background] Erickson KI, Colcombe SJ, Wadhwa R, Bherer L, Peterson MS, Scalf PE, Kim JS, Alvarado M, Kramer AF. Training-induced functional activation changes in dual-task processing: an FMRI study. Cereb Cortex. 2007 Jan;17(1):192-204. doi: 10.1093/cercor/bhj137. Epub 2006 Feb 8. PMID 16467562
- [Background] Eskelinen MH, Ngandu T, Helkala EL, Tuomilehto J, Nissinen A, Soininen H, Kivipelto M. Fat intake at midlife and cognitive impairment later in life: a population-based CAIDE study. Int J Geriatr Psychiatry. 2008 Jul;23(7):741-7. doi: 10.1002/gps.1969. PMID 18188871
- [Background] Friedman JI, Tang CY, de Haas HJ, Changchien L, Goliasch G, Dabas P, Wang V, Fayad ZA, Fuster V, Narula J. Brain imaging changes associated with risk factors for cardiovascular and cerebrovascular disease in asymptomatic patients. JACC Cardiovasc Imaging. 2014 Oct;7(10):1039-53. doi: 10.1016/j.jcmg.2014.06.014. PMID 25323165
- [Background] Hodyl NA, Schneider L, Vallence AM, Clow A, Ridding MC, Pitcher JB. The cortisol awakening response is associated with performance of a serial sequence reaction time task. Int J Psychophysiol. 2016 Feb;100:12-8. doi: 10.1016/j.ijpsycho.2015.12.007. Epub 2015 Dec 22. PMID 26721740
- [Background] Jennings JR, Muldoon MF, Ryan C, Price JC, Greer P, Sutton-Tyrrell K, van der Veen FM, Meltzer CC. Reduced cerebral blood flow response and compensation among patients with untreated hypertension. Neurology. 2005 Apr 26;64(8):1358-65. doi: 10.1212/01.WNL.0000158283.28251.3C. PMID 15851723
- [Background] Karssemeijer EGA, Aaronson JA, Bossers WJ, Smits T, Olde Rikkert MGM, Kessels RPC. Positive effects of combined cognitive and physical exercise training on cognitive function in older adults with mild cognitive impairment or dementia: A meta-analysis. Ageing Res Rev. 2017 Nov;40:75-83. doi: 10.1016/j.arr.2017.09.003. Epub 2017 Sep 12. PMID 28912076
- [Background] Kobe T, Witte AV, Schnelle A, Lesemann A, Fabian S, Tesky VA, Pantel J, Floel A. Combined omega-3 fatty acids, aerobic exercise and cognitive stimulation prevents decline in gray matter volume of the frontal, parietal and cingulate cortex in patients with mild cognitive impairment. Neuroimage. 2016 May 1;131:226-38. doi: 10.1016/j.neuroimage.2015.09.050. Epub 2015 Oct 1. PMID 26433119
- [Background] Launer LJ, Lewis CE, Schreiner PJ, Sidney S, Battapady H, Jacobs DR, Lim KO, D'Esposito M, Zhang Q, Reis J, Davatzikos C, Bryan RN. Vascular factors and multiple measures of early brain health: CARDIA brain MRI study. PLoS One. 2015 Mar 26;10(3):e0122138. doi: 10.1371/journal.pone.0122138. eCollection 2015. PMID 25812012
- [Background] Lupien SJ, Maheu F, Tu M, Fiocco A, Schramek TE. The effects of stress and stress hormones on human cognition: Implications for the field of brain and cognition. Brain Cogn. 2007 Dec;65(3):209-37. doi: 10.1016/j.bandc.2007.02.007. Epub 2007 Apr 26. PMID 17466428
- [Background] Lussier M, Gagnon C, Bherer L. An investigation of response and stimulus modality transfer effects after dual-task training in younger and older. Front Hum Neurosci. 2012 May 18;6:129. doi: 10.3389/fnhum.2012.00129. eCollection 2012. PMID 22629239
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Stampfer MJ, Hu FB, Manson JE, Rimm EB, Willett WC. Primary prevention of coronary heart disease in women through diet and lifestyle. N Engl J Med. 2000 Jul 6;343(1):16-22. doi: 10.1056/NEJM200007063430103. PMID 10882764
- [Background] van den Berg E, Kloppenborg RP, Kessels RP, Kappelle LJ, Biessels GJ. Type 2 diabetes mellitus, hypertension, dyslipidemia and obesity: A systematic comparison of their impact on cognition. Biochim Biophys Acta. 2009 May;1792(5):470-81. doi: 10.1016/j.bbadis.2008.09.004. Epub 2008 Sep 23. PMID 18848880
- [Background] Vianna LC, Deo SH, Jensen AK, Holwerda SW, Zimmerman MC, Fadel PJ. Impaired dynamic cerebral autoregulation at rest and during isometric exercise in type 2 diabetes patients. Am J Physiol Heart Circ Physiol. 2015 Apr 1;308(7):H681-7. doi: 10.1152/ajpheart.00343.2014. Epub 2015 Jan 16. PMID 25599569
- [Background] Wang R, Fratiglioni L, Laveskog A, Kalpouzos G, Ehrenkrona CH, Zhang Y, Bronge L, Wahlund LO, Backman L, Qiu C. Do cardiovascular risk factors explain the link between white matter hyperintensities and brain volumes in old age? A population-based study. Eur J Neurol. 2014 Aug;21(8):1076-1082. doi: 10.1111/ene.12319. Epub 2013 Dec 7. PMID 24313901
- [Background] Yamamoto N, Yamanaka G, Takasugi E, Ishikawa M, Yamanaka T, Murakami S, Hanafusa T, Matsubayashi K, Otsuka K. Lifestyle intervention reversed cognitive function in aged people with diabetes mellitus: two-year follow up. Diabetes Res Clin Pract. 2009 Sep;85(3):343-6. doi: 10.1016/j.diabres.2009.05.014. Epub 2009 Jun 10. PMID 19520452
- [Background] Zhu X, Yin S, Lang M, He R, Li J. The more the better? A meta-analysis on effects of combined cognitive and physical intervention on cognition in healthy older adults. Ageing Res Rev. 2016 Nov;31:67-79. doi: 10.1016/j.arr.2016.07.003. Epub 2016 Jul 14. PMID 27423932
- [Derived] Bherer L, Vrinceanu T, Dupuy EG, Gayda M, Vincent T, Magnan PO, Mohammadi H, Gauthier C, Gagnon C, Duchesne S, Erickson KI, Gagnon D, Lesage F, Lupien S, Poirier J, Dube MP, Thorin E, Juneau M, Breton J, Belleville S, Ferland G, Gaudreau-Majeau F, Blanchette CA, Vitali P, Nigam A. Investigating the effects of a randomized, double-blinded aerobic, resistance, and cognitive training clinical trial on neurocognitive function in older adults with cardiovascular risk factors: the ACTIONcardioRisk protocol. Front Aging Neurosci. 2025 Jun 23;17:1605128. doi: 10.3389/fnagi.2025.1605128. eCollection 2025. PMID 40625372